CLINICAL TRIAL: NCT01839604
Title: A Phase I/Ib, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of AZD9150 in Patients With Advanced/Metastatic Hepatocellular Carcinoma
Brief Title: A Phase I/Ib Study of AZD9150 (ISIS-STAT3Rx) in Patients With Advanced/Metastatic Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5660C00001; ISIS 481464 (Other: ISIS Pharmaceuticals Inc)
Record Dates: First submitted 2013-03-21; First posted 2013-04-25 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2016-05

CONDITIONS: Advanced Adult Hepatocellular Carcinoma; Hepatocellular Carcinoma Metastatic
Keywords: Child-Pugh A to B7,; Advanced/Metastatic Hepatocellular Carcinoma,; AZD9150,; Antisense Oligonucleotide Inhibitor of STAT3
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — danvatirsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD9150 (Experimental): There are two parts, dose escalation phase (Part A) and dose expansion phase (Part B).
  Interventions: Drug: AZD9150

INTERVENTIONS:
Drug: AZD9150 — Intravenous infusion over 3 hours.
  Other Names: ISIS 481464

SUMMARY:
This is a phase I/Ib open-label, multicentre study to assess the safety, tolerability, pharmacokinetics and preliminary anti-tumour activity of AZD9150 in patients with advanced/metastatic hepatocellular carcinoma.

DETAILED DESCRIPTION:
A Phase I/Ib, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of AZD9150 in Patients with Advanced/Metastatic Hepatocellular Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years. Patient from Japan and Taiwan aged at least 20 years
* Histologically or cytologically confirmed HCC (with the exception of fibrolamellar carcinoma or mixed variants of HCC with fibrolamellar histology OR clinically diagnosed HCC for patients with difficulty in obtaining histological diagnosis)
* Relapsed, refractory, intolerant or unlikely to benefit from sorafenib (for example due to comorbidity)
* Metastatic or locally advanced meeting ANY of the criteria below:
* HCC not suitable to receive local therapy
* Disease recurred or was refractory to last therapy (local or systemic)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 with no deterioration over the previous 2 weeks and minimum life expectancy of 8 weeks

Exclusion Criteria:

* More than 2 prior systemic treatments for HCC
* Prior grade 3 hematologic toxicity related to treatment with a JAK or STAT3 inhibitor
* Presence of hepatic encephalopathy within 4 weeks of 1st dose
* Uncontrolled massive ascites
* High likelihood of bleeding

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Neumann, MD, Study Director — AstraZeneca
Locations (7):
- Research Site, Hong Kong, Hong Kong
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Kashiwa-shi
  - Research Site, Matsuyama
- Research Site, Seoul, South Korea
- Taiwan (2):
  - Research Site, Tainan
  - Research Site, Taipei

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient entered the study on 03 May 2013, and the last patient last visit before the DCO was 31 December 2014. The DCO date was 05 January 2015.
Pre-assignment Details: Note that 39 patients is the number of patients who were actually assigned to treatment out of the total enrolled. The ecpansion phase consisted of the 3mg/kg group only.
Groups:
- AZD9150 1mg/kg: Intravenous. Part A.
- AZD9150 1.5 mg/kg; AZD9150 2mg/kg; AZD9150 2.5mg/kg: Intravenous dosing Part A
- AZD9150 3mg/kg: Pooled over parts A & B
Period: Overall Study
Arm/Group | AZD9150 1mg/kg | AZD9150 1.5 mg/kg | AZD9150 2mg/kg | AZD9150 2.5mg/kg | AZD9150 3mg/kg
Started | 6 | 6 | 7 | 5 | 15
Completed | 6 | 6 | 7 | 5 | 15
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1.5 mg/kg: given intravenously. Part A
- 2 mg/kg; 2.5 mg/kg: given intravenously Part A
- 3 mg/kg: given intravenously (Part A & B pooled)
- Total: Total of all reporting groups
Arm/Group | AZD9150 1mg/kg | 1.5 mg/kg | 2 mg/kg | 2.5 mg/kg | 3 mg/kg | Total
Number analyzed (Participants) | 6 | 6 | 7 | 5 | 15 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (13.0) | 58.3 (12.9) | 64.1 (10.4) | 58.0 (11.0) | 57.5 (8.9) | 59.2 (10.4)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 2 | 0 | 5
  Male | 6 | 5 | 5 | 3 | 15 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities During Cycle 1
Description: Cycle 1 was defined as 3 loading doses given on Days 1, 3, and 5 followed by 3 weekly doses given on Days 8, 15, and 22.
Time Frame: DLT assessment window - Cycle 1 (22 days)
Population: Safety: All patients who received at least 1 dose of AZD9150
Measure: Number; unit: participants with DLT
Arm/Group | AZD9150 1mg/kg | 1.5 mg/kg | 2 mg/kg | 2.5 mg/kg | 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 14
participants with DLT | 0 | 1 | 1 | 2 | 3

2. Secondary Outcome: Evaluation of Pharmacokinetics (PK) of AZD9150 (Following Single Administrations in Patients With HCC) by Determining Cmax, Using the Plasma Concentration Data.
Description: 8 times (pre-dose, 1.5, 3, 3.5, 4, 6, 8, 24 hours post-dose) on Day1 of Cycle1. For additional 6 patients in Japan, 8 times (pre-dose, 1.5, 3, 3.5, 4, 6, 8, 24 hours post-dose) on Day1 of Cycle1. From the multiple samples a timecourse is obtained of treatment conc in the plasma over time. From this curve the associated PK parameters e.g. Cmax are obtained. For n patients we obtain up to n parameters which can then be averaged.
Time Frame: 8 times of PK sampling on Day1 of Cycle1. Additional 6 patients in Japan; 8 times of PK sampling on Day1 of Cycle1.
Population: PK: All dosed patients with reportable AZD9150 plasma concentrations and no important adverse events or protocol deviations that may impact PK
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AZD9150 1mg/kg | 1.5 mg/kg | 2 mg/kg | 2.5 mg/kg | 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 7 | 5 | 15
ng/mL | 5833 (28.02) | 5575 (21.63) | 8984 (20.28) | 11560 (15.16) | 16110 (30.70)

3. Secondary Outcome: Preliminary Assessment of the Anti-tumour Activity of AZD9150 by Evaluation of Tumour Response.
Description: Tumour response assessment by modified Response Evaluation Criteria in Solid Tumours (RECIST). Overall tumour response: assessed by mRECIST for HCC overall visit response of CR (disappearance of baseline TLs and NTLs), PR (>=30% decrease in sum of TLs), SD (neither PR nor PD), PD (sum TLs increased >20%), or NE .
Time Frame: Every 6 weeks, assessed up to 12 months.
Population: Evaluable for response: Dosed patients with measurable disease at baseline
Measure: Number; unit: participants with Partial Response
Arm/Group | AZD9150 1mg/kg | 1.5 mg/kg | 2 mg/kg | 2.5 mg/kg | 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 7 | 5 | 15
participants with Partial Response | 0 | 0 | 1 | 0 | 0

4. Secondary Outcome: Evaluation of Pharmacokinetics (PK) of AZD9150 (Following Single Administrations in Patients With HCC) by Determining Tmax, Using the Plasma Concentration Data.
Description: 8 times (pre-dose, 1.5, 3, 3.5, 4, 6, 8, 24 hours post-dose) on Day1 of Cycle1. For additional 6 patients in Japan, 8 times (pre-dose, 1.5, 3, 3.5, 4, 6, 8, 24 hours post-dose) on Day1 of Cycle1.
Time Frame: 8 times of PK sampling on Day1 of Cycle1. Additional 6 patients in Japan; 8 times of PK sampling on Day 1 of Cycle 1.
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | AZD9150 1mg/kg | 1.5 mg/kg | 2 mg/kg | 2.5 mg/kg | 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 7 | 5 | 15
h | 3.0 [1.5 to 3.0] | 3.4 [3.0 to 3.7] | 2.8 [1.5 to 3.5] | 3.0 [2.9 to 3.5] | 3.0 [1.3 to 3.0]

ADVERSE EVENTS:
Time Frame: AEs will be collected throughout the study, from informed consent until the end of the follow up period. The follow-up period is defined as 28 +/-7 days after study treatment is discontinued.
Arm/Group | AZD9150 1mg/kg | 1.5 mg/kg | 2 mg/kg | 2.5 mg/kg | 3 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 2/7 | 2/5 | 4/15
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 7/7 | 5/5 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9150 1mg/kg (N=6) | 1.5 mg/kg (N=6) | 2 mg/kg (N=7) | 2.5 mg/kg (N=5) | 3 mg/kg (N=15)
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1)
Liver abscess (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 (1) | 0 (0)
Alanine amonitransferase increased (Investigations) | 0 | 0 | 1 (1) | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 (1) | 1 (1) | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 (1)
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9150 1mg/kg (N=6) | 1.5 mg/kg (N=6) | 2 mg/kg (N=7) | 2.5 mg/kg (N=5) | 3 mg/kg (N=15)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 4 (4) | 5 (5) | 3 (3) | 9 (9)
Platelet count decreased (Investigations) | 3 (3) | 3 (3) | 5 (5) | 1 (1) | 10 (10)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (3) | 4 (4) | 3 (3) | 9 (9)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gamma-glutamylytransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
White blod cell count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 2 (2) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 (2) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 1 (1) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 1 (1) | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 1 (1) | 0
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 | 2 (2) | 0 | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 1 (1) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0 | 2 (2)
Fatigue (General disorders) | 0 | 0 | 0 | 1 (1) | 3 (3)
Pyrexia (General disorders) | 0 | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 | 1 (1) | 1 (1) | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Decreased apetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 1 (1) | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The overall study objectives were achieved earlier than anticipated, so recruitment was stopped and the study was considered complete. In turn multiple dose PK profiles were not obtained during the study expansion phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less